CLINICAL TRIAL: NCT05345639
Title: Chest Wall Block After Sternotomy: Randomized Controlled Trial in Cardiac Surgery: (PABLOS Study)
Acronym: PABLOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49RC21_0251
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-12

CONDITIONS: Pain, Postoperative; Cardiac Surgery
Keywords: LRA; Block; ERAS; FQOR-15; QOR-15; Transversus thoracic block; Parasternal block; Cardiac surgery; Analgesia; PIP (parasternal intercostal plane block); Régional anesthesia
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings; Agnosia

STUDY DESIGN:
Intervention Model Description: Study phase III, superiority study, monocentric, comparative, with three parallel groups, randomized with a ratio (1:1:1), controlled versus standard care, single-blind
Who Masked: Participant
Masking Description: Randomization takes place during surgery. Bilateral parasternal block or transverse thoracic block are performed ultrasound-guided, under general anesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TTP group (= Transversus Thoracic Plane block = Deep PIP = Deep parasternal intercostal plane block) (Experimental): At the end of the surgery, realisation of a bilateral transverse thoracic block. (20ml of Naropeine 0.2%, each side) Followed by standard analgesic treatment.
  Interventions: Drug: LRA Loco-regional anesthesia; Procedure: Standardized post-operative analgesia protocol
- PSB group (=ParaSternal Block = Superficial PIP = Superficial parasternal intercostal plane block) (Experimental): At the end of the surgery, realisation of a bilateral parasternal block (20ml of Naropeine 0.2%, each side).
  Followed by standard analgesic treatment.
  Interventions: Drug: LRA Loco-regional anesthesia; Procedure: Standardized post-operative analgesia protocol
- Control group (Sham Comparator): Standard analgesic treatment alone (without LRA) .
  Interventions: Procedure: Standardized post-operative analgesia protocol

INTERVENTIONS:
Drug: LRA Loco-regional anesthesia — Bilateral parasternal block or transverse thoracic block are performed ultrasound-guided, at the end of surgery in the operating room. Once in the desired plane depending on the randomisation (transverse or parasternal), a volume of 20 ml of ropivacaine at 2 mg/ml is injected on each side of the sternum.
  The intervention (TTP or PSB) is performed by the anesthetist-resuscitator investigator.
  Other Names: 40ml Ropivacaine 0.2%
  Arms: PSB group (=ParaSternal Block = Superficial PIP = Superficial parasternal intercostal plane block); TTP group (= Transversus Thoracic Plane block = Deep PIP = Deep parasternal intercostal plane block)
Procedure: Standardized post-operative analgesia protocol — The pain management protocol in intensive care is as follows:
  * paracetamol 1g x 4 per day systematically (apart from the usual contraindications), IV then PO;
  * PCA (Patient Controlled Analgesia) with oxycodone or morphine: 1mg bolus, 7min refractory period, maximum 4h dose 20mg.
  The PCA is usually maintained until 24-48h after the intervention then relayed by oxycodone 5mg every 4h if EVA > 3 sublingual and addition of oxycodone LP 10mg x 2 per day if daily intake on PCA > 20mg.
  Remedy molecules in case of ineffective analgesia:
  ketoprofen 100mg q12h IV, or 50mg q8h PO; nefopam 20mg every 6h IV or PO; ketamine 1 to 1.5 mg/kg/24H IVSE.

SUMMARY:
The main objective is to compare the effectiveness of LocoRegional Anesthesia (LRA) (bilateral transverse thoracic block or bilateral parasternal block) in addition to standard management compared to standard management alone (general anesthesia without LRA) on the FQoR-15 (French Quality of Recovery - 15 score) at H+24 after cardiac surgery by sternotomy.This is a phase III monocentric superiority study , comparative, with three parallel groups, randomized with a ratio (1:1:1), controlled versus standard management, single-blind.

DETAILED DESCRIPTION:
Each year, more than one million patients worldwide undergo cardiac surgery via sternotomy. Postoperative pain is frequent in this context, affecting 49% of patients at rest and 78% during mobilization. This pain is associated with many avoidable post-operative complications.

Nowadays, ERAS (Enhanced Rehabilitation After Surgery) protocols are increasingly developed in order to optimize post-operative rehabilitation. The management of postoperative pain is one of their main challenges and is based in particular on the use of locoregional anesthesia (LRA) with the aim of sparing morphine.

Several LRAs have been described in cardiac surgery in recent years, and they are increasingly used in routine clinical practice. Transverse thoracic block and parasternal block are the main peripheral LRA techniques proposed for surgical procedures with sternotomy. Transverse chest block was first described in cardiac surgery in 2015 ; and the parasternal block in 2018. These techniques are spreading in current clinical practice because of their simplicity of implementation, their safety and their supposed effectiveness. The parasternal block is more recent, and presents a more superficial injection plane than the transverse thoracic block. Thus, it is theoretically as effective as the transverse thoracic and less at risk of complications.

The main objective of this study is to compare the effectiveness of LRA (bilateral transverse thoracic block or bilateral parasternal block) in addition to standard management compared to standard management alone (general anesthesia without LRA) on the quality of early postoperative recovery after heart surgery by sternotomy.

The primary endpoint is the postoperative recovery score in the French version, FQoR-15 (French Quality of Recovery - 15 score), performed at H+24. The FQoR-15 is currently one of the most reliable and reproducible tools for assessing the quality of postoperative rehabilitation. This instrument is one of the recommended endpoints for the evaluation of patient comfort, according to a recent consensus of international experts.

This study is a phase III study of superiority, monocentric, comparative, with three parallel groups, randomized with a ratio (1:1:1), controlled versus standard care, single-blind. of inclusion is 254 patients included and randomized.

The patient is pre-included during the pre-anaesthetic visit, the day before his scheduled surgery. He receives oral and written information, and provides his written consent to participate in this study, the follow-up will be 30 days. Depending on the randomization, the patient receives one of the following three treatments:

1. bilateral transverse thoracic block followed by standard analgesic management;
2. a bilateral parasternal block followed by standard analgesic treatment;
3. standard analgesic treatment alone (without LRA). Bilateral parasternal block or transverse thoracic block are performed ultrasound-guided, at the end of surgery in the operating room. Once in the desired plane depending on the randomisation (transverse or parasternal), a volume of 20 ml of ropivacaine at 2 mg/ml is injected on each side of the sternum. The rest of the pain management is identical in the three groups according to the habits of the department.

If the hypotheses on the effectiveness of parasternal block and/or transverse thoracic block are confirmed, postoperative recovery in the interventional arms will be improved. This will confirm the value of performing an LRA postoperatively.

ELIGIBILITY:
Pre-inclusion criteria :

* Adult patient (≥18 years old);
* Patient having scheduled cardiac surgery with a sternotomy performed at the CHU d'Angers;
* Patient having signed a consent;
* French-speaking patient, able to understand and answer a questionnaire;
* Affiliated patient or beneficiary of a social security scheme.

Criteria for confirming inclusion

* Hemodynamic stability at the end of surgery;
* Absence of bleeding justifying immediate revision surgery.

Non-inclusion criteria

* Known hypersensitivity to amide-bonded local anesthetics;
* Operation for cardiac revision surgery, including sternotomy REDUX (revision surgery);
* Emergency surgery;
* Surgery in a septic context (Endocarditis, Intravascular device infection);
* Weight less than 30kg;
* Severe psychiatric or cognitive impairment interfering with assessment by questionnaires;
* Pregnant, breastfeeding or parturient woman;
* Person deprived of liberty by judicial or administrative decision;
* A person undergoing psychiatric treatment under duress;
* Person subject to a measure of legal protection;
* Inclusion in another interventional study modifying postoperative pain management.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
FQoR-15 score at 24 hours (French Quality of Recovery-15 score) | 24 hours after surgery
  Value of the French Quality of Recovery-15 score (minimum value of 0 and maximum value of 150, with a higher score for a better outcome).
  The QoR-15 questionnaires will be completed by the patient himself whenever possible, who could be helped by a nurse blinded to the assignment group.

SECONDARY OUTCOMES:
Pain (VRS) at rest and mobilisation | 3, 6, 12, 24, 48 , 72 hours after surgery and during the removal of surgical drains
  Analgesic efficacy at rest and during exercise (cough, physiotherapy session, mobilization) assessed via pain measurements by a simple verbal rating scale (VRS) with 11 items (0: no pain, 10: maximum pain)
Post-operative consumption of morphine (milligrams) | 3, 6, 12 hours after surgery and daily assessed at 24, 48, 72, 96 and 120 hours after surgery
  Amount of opioid consumption, in equivalent of milligrams.
Post-operative consumption of daily non-morphine analgesics (milligrams) | 24, 48, 72, 96 and 120 hours after surgery
  Including Pacetamol, Nefopam, ketoprofene, Ketamine in milligrams.
Rate of painful patients | 24 and 48 hours after surgery
  Proportion of patients having had at least one VRS >3
FQoR-15 score at 48 hours | 48 hours after surgery
  The quality of postoperative recovery reassessed 48 hours after surgery by the FQoR-15; Value of the French Quality of Recovery-15 score (minimum value of 0 and maximum value of 150, with a higher score for a better outcome).
  The QoR-15 questionnaires will be completed by the patient himself whenever possible, who could be helped by a nurse blinded to the assignment group.
Rate of patients with at least one complication of LRA | 30 days
  Proportion of patients with at least one complication of LRA: systemic intoxication with local anesthetics within 3 hours after injection, hematoma or infection at the puncture site.
Rate of postoperative complications | 30 days
  The proportion of patients with at least one major postoperative complication of cardiac surgery during hospitalization: de novo postoperative atrial fibrillation, revision surgery, respiratory failure, mediastinitis, neurological complication, acute renal failure, gastrointestinal complication, infectious complication with bacteremia, pneumothorax, infectious pneumonitis.
Rate of patients return to preoperative weight | Noted at day 3 and 5 after surgery
  Proportion of patient return to announced weight at the pre-anaesthetic consultation (truncating the weight in kg)
Rate of patients return to a transit | Noted at day 3 and 5 after surgery
  Proportion of patient return to a transit (including solid or gaseous transit)
Extubation time (hours) | Noted at Day 30
  Measured in number of hours since arrival in intensive care (between arrival in intensive care and the first attempt at extubation);
Duration of hospitalization. (days) | Noted at Day 30
  The length of stay in post-operative intensive care (between arrival in intensive care and leaving the service) and in the hospital counted in number of days started.
Rate of readmission to intensive care. | Noted at Day 30
  The proportion of patients admitted in the intensive care unit whatever the reason, censored at 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Jeanneteau, Angers, maine et loire, France

IPD SHARING:
Plan to Share IPD: No
The data will be collected in a coded manner: 1st letter of the surname, 1st letter of the patient's first name, serial number of inclusion in the center by the physicians investigating the study in the electronic observation notebook of the study ( EnnovClinical) managed by the DRCI of the CHU of Angers.

REFERENCES:
- [Background] Bignami E, Castella A, Pota V, Saglietti F, Scognamiglio A, Trumello C, Pace MC, Allegri M. Perioperative pain management in cardiac surgery: a systematic review. Minerva Anestesiol. 2018 Apr;84(4):488-503. doi: 10.23736/S0375-9393.17.12142-5. Epub 2017 Oct 12. PMID 29027773
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Background] Huang AP, Sakata RK. Pain after sternotomy - review. Braz J Anesthesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjane.2014.09.013. Epub 2016 Apr 23. PMID 27343790
- [Background] McIsaac DI, Cole ET, McCartney CJ. Impact of including regional anaesthesia in enhanced recovery protocols: a scoping review. Br J Anaesth. 2015 Dec;115 Suppl 2:ii46-56. doi: 10.1093/bja/aev376. PMID 26658201
- [Background] Ueshima H, Hara E, Marui T, Otake H. RETRACTED: The ultrasound-guided transversus thoracic muscle plane block is effective for the median sternotomy. J Clin Anesth. 2016 Mar;29:83. doi: 10.1016/j.jclinane.2015.10.014. Epub 2016 Feb 9. No abstract available. PMID 26897453
- [Background] de la Torre PA, Garcia PD, Alvarez SL, Miguel FJ, Perez MF. A novel ultrasound-guided block: a promising alternative for breast analgesia. Aesthet Surg J. 2014 Jan 1;34(1):198-200. doi: 10.1177/1090820X13515902. No abstract available. PMID 24396082
- [Background] Leger M, Campfort M, Cayla C, Parot-Schinkel E, Lasocki S, Rineau E. Validation of an alternative French version of the Quality of Recovery-15 Score: the FQoR-15. Br J Anaesth. 2020 Oct;125(4):e345-e347. doi: 10.1016/j.bja.2020.05.052. Epub 2020 Jul 9. No abstract available. PMID 32654751
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Myles PS, Boney O, Botti M, Cyna AM, Gan TJ, Jensen MP, Kehlet H, Kurz A, De Oliveira GS Jr, Peyton P, Sessler DI, Tramer MR, Wu CL; StEP-COMPAC Group; Myles P, Grocott M, Biccard B, Blazeby J, Boney O, Chan M, Diouf E, Fleisher L, Kalkman C, Kurz A, Moonesinghe R, Wijeysundera D. Systematic review and consensus definitions for the Standardised Endpoints in Perioperative Medicine (StEP) initiative: patient comfort. Br J Anaesth. 2018 Apr;120(4):705-711. doi: 10.1016/j.bja.2017.12.037. Epub 2018 Feb 2. PMID 29576111
- [Derived] Demarquette A, Jeanneteau A, Blanchard-Daguet A, Fouquet O, Parot-Schinkel E, Lasocki S, Rineau E, Leger M. Impact of superficial and deep parasternal blocks on recovery after cardiac surgery with sternotomy: a randomised controlled trial. Br J Anaesth. 2025 Sep;135(3):764-771. doi: 10.1016/j.bja.2025.05.043. Epub 2025 Jul 9. PMID 40640047
- [Derived] Jeanneteau A, Demarquette A, Blanchard-Daguet A, Fouquet O, Lasocki S, Riou J, Rineau E, Leger M. Effect of superficial and deep parasternal blocks on recovery after cardiac surgery: study protocol for a randomized controlled trial. Trials. 2023 Jul 6;24(1):444. doi: 10.1186/s13063-023-07446-2. PMID 37415221